CLINICAL TRIAL: NCT02299778
Title: Is Bacterially-Synthesized Folate Absorbed Across the Colon of Humans?
Brief Title: Bacterially-synthesized Folate Absorption Across the Large Intestine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Deborah O'Connor, Senior Associate Scienitst, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1000026022
Record Dates: First submitted 2014-10-23; First posted 2014-11-24 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1mg of 13C6-p-aminobenzoic acid (Experimental)
  Interventions: Dietary Supplement: 13C6-p-aminobenzoic acid

INTERVENTIONS:
Dietary Supplement: 13C6-p-aminobenzoic acid

SUMMARY:
The purpose of this study is to determine whether folate produced by bacteria that live in our colon can be absorbed in human colon using a stable isotope method. This study would lead a better understanding of the bioavailability of colonic bacterially-synthesized folate and its quantitative contribution to whole body folate homeostasis.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years;
2. overall healthy

Exclusion Criteria:

1. <18 years or >65 years
2. chronic disease (eg. history of hepatic, gastrointestinal, renal, vascular, haematological or neuropsychiatric disease) or surgery affecting gastrointestinal motility, pH or folate absorption/metabolism
3. regular use of medications affecting gastrointestinal pH, motility or folate absorption/metabolism (eg. antiacids, laxatives, phenytoin, sulfasalzine, phenobarbital, primidone, cimetidine, proton pump inhibitors [such as Nexium] and antibiotics [such as Sulfonamides] or nonsteroidal anti-inflammatory drugs [NSAIDS, such as aspirin/ibuprofen])
4. consumption of >1 drink/day of alcohol on a regular basis or current smoking (last 6 months)
5. planning a pregnancy, pregnant, breast feeding or the use of high-dose estrogen oral contraceptives/hormone replacement therapy
6. known sensitivity to sunscreens containing ultraviolet B filters and/or PABA
7. difficulty with swallowing large pills or providing venous blood samples

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in isotopic folate overtime in blood | Baseline (day 1), Days 2-4 ( 0h,1h,2h,3h,4h,5h,6h,7h,8h,9h,10h,11h,12h,24hr,48hr)
Change in isotopic folate overtime in urine | Day 1 (0-24hr), Day 2 (25-48hr), Day 3 ( 49-72hr), Day 4 (73-96hr)

SECONDARY OUTCOMES:
Folate intake | Day1-4
  Assessed using food records
Fiber intake | Day1-4
  Assessed using food records

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L O'Connor, RD, PhD, Principal Investigator — The Hospital for Sick Children, Toronto, ON, Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada